CLINICAL TRIAL: NCT05091476
Title: A Clinical Study to Evaluate the Safety and Feasibility of the OcuDyne System in the Treatment of Age-Related Macular Degeneration (AMD)
Brief Title: OcuDyne System in the Treatment of AMD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OcuDyne, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OC-1901AR
Record Dates: First submitted 2021-10-12; First posted 2021-10-25 (Actual); Last update posted 2025-02-13 (Actual); Status verified 2025-02

CONDITIONS: Age-Related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Eyes treated with the OPTiC System (Experimental): Eyes that OPTiC System treatment has been completed
  Interventions: Device: OPTiC System
- Fellow Eye (No Intervention): Contralateral comparator

INTERVENTIONS:
Device: OPTiC System — OPTiC System procedure
  Arms: Eyes treated with the OPTiC System

SUMMARY:
Feasibility of the OcuDyne OPTiC System in patients with late-stage non-exudative age-related macular degeneration.

DETAILED DESCRIPTION:
This study evaluates the safety and feasibility of using the OcuDyne OPTiC System in patients with late-stage non-exudative age-related macular degeneration.

ELIGIBILITY:
Inclusion Criteria:

1. Must be able to understand and provide informed consent on an Independent Ethics Committee (EC) approved informed consent form (ICF)
2. Must be willing and able to return for scheduled treatment and follow-up examinations for up to a 7-month duration
3. Adults at least 60 years of age at the time of consent
4. Diagnosed with non-exudative Age-Related Macular Degeneration with current or previous evidence of at least one large drusen (measuring 125 microns or greater) and nascent geographic atrophy (nGA) or GA in the study eye
5. ETDRS best corrected visual acuity (BCVA) letter score of less than 56 letters (Snellen equivalent of 20/80 or worse) in the study eye, which in the Investigator's judgment is caused by non-exudative age-related macular degeneration (AMD)
6. The confirmed presence of ophthalmic artery (OA) stenosis (leading to the study eye).

Exclusion Criteria:

OCULAR

1. Any surgical intraocular treatment (including laser) within 3 months in the study eye.
2. History of exudative AMD or Anti-Vascular Endothelial Growth Factor (anti-VEGF) injections within 6 months in the study eye.
3. Presence of ocular media affecting visual acuity or the ability to visualize the retina in either eye (e.g., central corneal scarring, lens opacities along visual axis, posterior capsule opacification, etc.).
4. History of chronic, recurring inflammatory eye disease in either eye (e.g., scleritis, uveitis, corneal edema, etc.)
5. Presence of diabetic retinopathy in either eye.
6. Evidence of macular edema secondary to exudation in the study eye.
7. History of amaurosis fugax, central or retinal artery or vein occlusion, anterior ischemic optic neuropathy (AION) or non-arteritic anterior ischemic optic neuropathy (NAION) or any diagnosis of a macular disease other than AMD such as Stargardt disease, cone rod dystrophy, angioid streaks, or toxic maculopathies such as Plaquenil maculopathy.
8. Myopia > 6.0 Diopters (D) spherical equivalent (SE) or Axial Length ≥ 26.0 mm in the study eye.
9. Presence of visually significant epiretinal membrane in the study eye.
10. Participation in any eye-related drug or device clinical trial involving either eye within 90 days prior to enrolling in this study and/or during study participation.

    Non-Ocular
11. Any condition that prohibits the use of intravenous contrast agents (e.g., renal insufficiency, previous anaphylactoid reaction to contrast material, treatment with nephrotoxic agents, etc.).
12. Previous stroke, including ischemic, hemorrhagic or transient ischemic attack (TIA).
13. Previous myocardial infarction (MI), including ST segment elevation (STEMI), non-ST segment elevation (NSTEMI) or coronary spasm/angina.
14. Coronary or other intravascular percutaneous procedure, including balloon angioplasty, stent or filter placement within the last 6 months.
15. Complete occlusion of the ophthalmic artery.
16. Pacemaker, Cochlear, or neurostimulation implant.
17. Presence of cranial aneurysm, clinically significant stenosis in common carotid artery or internal carotid artery, or tortuous vascular anatomy as seen on pre-procedural CT Angiogram that, in the clinical judgement of the investigator, represents an unreasonable risk to perform the intervention.
18. Condition associated with increased bleeding risk including but not limited to: major surgical procedure or trauma within 30 days of screening; clinically significant gastrointestinal bleeding within 1 year of screening; known gastric or duodenal ulcer; history of intracranial or spinal bleeding; chronic hemorrhagic disorder; treatment with oral anticoagulant medications (e.g., Warfarin / non-vitamin K anticoagulants [NOACs] exclusionary; aspirin or clopidogrel allowed), known intracranial neoplasm, arteriovenous malformation, or aneurysm.
19. Treatment with oral anticoagulant medications (e.g., Warfarin / non-vitamin K anticoagulants [NOACs] exclusionary; aspirin or clopidogrel allowed).
20. Sustained and uncontrolled hypertension with systolic blood pressure > 180 mmHg.
21. Diagnosis of moderate to severe symptomatic congestive heart failure (CHF) or chronic obstructive pulmonary disease (COPD)
22. Diagnosis of connective tissue, demyelinating, autoimmune, or inflammatory diseases (e.g., lupus, rheumatoid arthritis, scleroderma, giant cell arteritis, multiple sclerosis, etc.).
23. Intolerance of either pre- or post- procedure medication regimen.
24. Pregnancy, lactation, or plans to become pregnant during participation in this clinical trial.
25. Participation in any other non-eye related drug or device clinical trial within 30 days prior to enrolling in this study and/or during study participation.

    Other
26. Use of facial fillers or paralytic drugs during study participation.
27. Subject who, in the clinical judgement of the investigator, is not otherwise suitable for participation in the study for another clinical reason, as documented by the investigator.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2023-02-27 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Adverse Events | Intraoperative through Week 4 postoperative
  Procedural Complications & Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Luana R Wilbur, BS, Study Director — OcuDyne VP, Clinical and Regulatory Affairs
Locations (2):
- Argentina (2):
  - Buenos Aires Macula, Buenos Aires
  - ENERI, Buenos Aires

IPD SHARING:
Plan to Share IPD: No